CLINICAL TRIAL: NCT05142007
Title: The Effect of Hypnotic Suggestion on Return to Work, Functioning, and Cognition Following Acquired Brain Injury or Concussion: A Randomized Controlled Trial
Brief Title: The Effect of Hypnotic Suggestion After Acquired Brain Injury or Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Defactum, Central Denmark Region (Other Government)
Responsible Party: Principal Investigator, Pernille Pedersen, Senior researcher, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 342096
Record Dates: First submitted 2021-10-29; First posted 2021-12-02 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Acquired Brain Injury; Concussion, Brain
Keywords: Brain Injuries; Brain Concussion; Hypnosis; Return To Work; Sick Leave; Randomized Controlled Trial [Publication Type]
MeSH Terms: conditions — Brain Injuries; Brain Concussion | interventions — Hypnosis; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (Experimental): The first treatment arm ("targeted suggestion") consist of suggestions about enhancing working memory functions through the instantiation of preinjury working memory ability in the present using age regression, visualizations of neuroplasticity in the present, and posthypnotic suggestions about continued improvement. The overarching theme of the suggestions is that thinking itself will become effortless and reliable, leading to reduced fatigue, better memory, and the absence of information overload.
  Interventions: Behavioral: Hypnosis
- Mindfulness-based stress reduction (Active Comparator): The second treatment arm ("non-targeted suggestion" or MBSR) contains no explicit mentioning of brain injury or working memory-related abilities and thus serves to isolate the 'targetedness' of suggestion as well as factoring out other influences from placebo, retest effects, etc.
  Interventions: Behavioral: Mindfulness-based stress reduction
- Control group (No Intervention): The (passive) control group receives no contact over and beyond testing.

INTERVENTIONS:
Behavioral: Hypnosis — A number of steps are taken to make the treatment arms identical in all other respects. The participants are unaware that there are two treatment arms to homogenize expectations. Each session is a manualized hypnosis script which is dictated by the hypnotist, including the hypnosis test. The only degrees of freedom for the hypnotist is in intonation and speed. Identical induction and termination is used in both arms and the scripts are of comparable durations.
  Arms: Hypnosis
Behavioral: Mindfulness-based stress reduction — A number of steps are taken to make the treatment arms identical in all other respects. The participants are unaware that there are two treatment arms to homogenize expectations. Each session is a manualized hypnosis script which is dictated by the hypnotist, including the hypnosis test. The only degrees of freedom for the hypnotist is in intonation and speed. Identical induction and termination is used in both arms and the scripts are of comparable durations.
  Arms: Mindfulness-based stress reduction

SUMMARY:
A recent randomized clinical trial (RCT) demonstrated large effects of hypnotic suggestion on working memory following acquired brain injury. However, no studies have investigated long-term effects (> 2 months) effects on return to work (RTW).

Therefore the aim is in a RCT to study the effect of hypnotic suggestion on RTW in employed individuals with acquired brain injury or concussion, that were referred to an out-patient municipal vocational rehabilitation center in Denmark.

Participants were randomized to a passive (treatment as usual), active comparison (a weekly treatment session of mindfullness-based stress reduction for four weeks) or intervention group (a weekly treatment session of targeted suggestion for four weeks).

Intention-to-treat analysis of the hypnosis effect on return to work within six months follow-up will be performed.

Results Participants (N=77) have accepted and participated in the study. Effect measures are to be analysed.

DETAILED DESCRIPTION:
Introduction Hypnotic suggestion may be an effective treatment modality for cognitive sequelae following acquired brain injury and concussion. A recent RCT demonstrated large effects of hypnotic suggestion on working memory following acquired brain injury. Analyses of interview-data from that RCT also indicated large effects on sleep and Patient-Reported Outcomes (PROs). Previous studies have similarly shown clinically notable effects in the cognitive domain, although these have some methodological shortcomings. While stroke and concussion patients exhibit non-impaired responsiveness to hypnotic suggestion, there is little literature on the effect of hypnotic suggestion on concussion patients. In a non-controlled study, it was found that vertigo was completely removed following 1-10 sessions of hypnosis in 63 out of 108 concussed patients and that vertigo was reduced in further 17 patients leaving only 28 (one in four) with no effect. In another smaller non-controlled study on patients with Mild Traumatic Brain Injury (MTBI), large effects on fatigue, anxiety, and depression were found. While the investigators have speculated about the mechanisms underlying the effect, the current goal of this research program is to provide the empirical basis for a verdict on whether hypnotic suggestion can be recommended for clinical practice. This is a pressing issue since brain injuries (stroke and TBI) constitute the world's second-most expensive health-related disability.

Long-term effects on everyday outcome measures is of utmost importance in clinical settings. However, no studies have investigated long-term (> 2 months) effects on Return to Work, participation in society, or fatigue, and only one high-quality RCT has been conducted. Here, the investigators present the protocol for an RCT that aims to fill in these gaps. The present protocol is an effectiveness study in a vocational-rehabilitation setting, but in other respects, it closely replicates the efficacy study by the primary investigator.

Objectives Estimate the effect of hypnotic suggestion on short- and long-term effects on Return to Work, participation in society, fatigue, and cognition. Given the promising findings in previous studies, the investigators hypothesize that hypnotic suggestion has positive effects in each of these domains.

Methods (setting) All patient activities take place at an out-patient municipal vocational rehabilitation center in Denmark, including recruitment, testing, and treatment. The center specifically offers support to increase labor market attachment.

Methods (recruitment) Potential participants were recruited from two departments in the vocational rehabilitation center: (1) a department specializing in citizens with brain-injury, concussion, whiplash, and related conditions. (2) A more general department which serviced a high rate of participants who had suffered a concussion. In both departments, the staff handed out participant information materials to all citizens who met inclusion 1-3 (age, etiology, and vocational history). The participants could optionally consent to giving their contact details to the project, contact the project by themselves, or decline. The first point of contact with the project was an oral information. The participant was given three days to consider consenting, though all participants made the decision immediately. After an initial screening by a project assistant, a list of eligible participants was sent to a dedicated non-blinded "coordinator" who randomly assigned participants to the groups while monitoring the balance between groups.

Methods (Sequence generation)

The coordinator used a computerized random sequence generator to assign participants to the three intervention groups. A practical constraint (unknown by the testers) was that a hypnotist should have exactly 5 participants in a day, if any. The procedure for randomization was:

When there were 5+ screened participants, assign random numbers to the participants and allocate the participants with the lowest 5 numbers to a "general intervention group" and the rest to the passive control group. Then assign new random numbers to the intervention-allocated participants and assign the participants with the lowest N numbers to SBCR and the others to mindfulness. N is the number that would make the two intervention groups equal in size in the full dataset.

If the number of passive controls exceeded the intervention groups, allocate 10 participants to the "general intervention group" and proceed cf. above. If the number of passive controls lacked the number in each intervention group, assign all participants to the passive control condition.

Methods (Implementation and blinding) A dedicated project assistant (the "coordinator") allocated participants, informed them of their allocation, and booked a hypnotist. The participants only knew that there was a "hypnosis" and a "control" group but were blind to the fact that there were, in fact, two hypnosis groups. Participants were encouraged to only disclose their allocation with close peers that were not at the vocational center. The testers, center staff, principal investigator, data analysts, and other professionals were unaware of the allocation throughout the study.

The allocation was saved at a secure server which only the coordinator had access to. The blinding was lifted when the last participant had had the 6-month follow-up test.

The coordinator and hypnotists were unaware of the testing results. Participants were given a brief overview of their testing results upon completion of the 6-months follow-up.

Blinding could be lifted for a single participant in case of serious side effects. If the side effect was serious enough to warrant halting the study, all blinding would be lifted to identify at-risk participants. The participants reported no serious side effects, so this procedure was never exercised.

Methods (Data management) All questionnaire data were entered electronically to ensure data quality and completeness. Computerized tests were saved in csv files by the program. In-person administered tests were recorded in dedicated scoring sheets and then entered digitally. The testers saved all screening- and outcome data to a secure server, which only the testers had access to.

Methods (Analysis) Intention-to-treat analysis of the hypnosis effect on return to work within six months' follow-up will be performed. The statistical software package Stata will be used.

Ethics The study was approved by the regional ethics committee (The North Denmark Region), journal number N-20170022. Any participant-facing changes to the study were approved there. Participants always completed on the protocol they started.

The consent was collected by the tester role in the "screening" section of the participant flow. The participant received written participant information in advance and an in-person oral information which briefly repeated the written materials and opened for discussion. Participants were given three days to consider whether to consent, though all participants decided immediately. The written consent was stored in a locker to which only testers had access.

Declaration of interest The authors declare no financial interest in the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented concussion or acquired brain injury which is at least 6 months old at the first (potential) therapy session.
* Employment more than 50% of the time after finishing the latest education and employed at least 6 consecutive months immediately preceding the injury
* If the patient is currently fully employed, he/she must have substantial risk of decreasing vocational status.
* No substance abuse or issues currently in- or requiring- psychiatric treatment.

Exclusion Criteria:

* Progressive injuries are excluded, including dementias.
* Pensioned or recommended for pension at the time of inclusion,

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Return to work | Within one year of follow-up
  The probability of returning to work is based on registry-based data. Dichotomous outcome: 0 (no), 1 (yes).

SECONDARY OUTCOMES:
WAIS-IV Working Memory Index | Six months follow-up
  Range of outcome: 50 (worst) to 150 (best). Age-corrected index computed from the performance on three tasks: mental arithmetic, letter span, and letter-number sequencing. They are scored, aggregated, and converted to index scores according to the WAIS-IV manual (Wechsler, 2008). Briefly, the manual contains tables where raw scores are converted to age-corrected scaled scores, the sum of which corresponds to an index value.
Trail Making Test (executive component of working memory) | Six months follow-up
  Trail Making Test is scored by how long it takes to complete the test (max 5 minutes). Executive task switching is assessed using the log(B-A) index of the Trail Making Task form A and B. Range of outcome: -Infinity (worst) to +Infinity (best) log-seconds with expected values in the range [0, 4] log-seconds.
  The outcome is the log-difference score between reaction times (outcome = log(B - A)).
Go-nogo reaction time difference | Six months follow-up
  Executive inhibition is assessed as go-nogo reaction time minus simple reaction time.
  Range of outcome: The difference score between simple reaction time and discrimination time (complex reaction time). From -Infinity (best) to Infinity (worst) with expected mean differences in the range [0.1, 0.5], [best, worst]seconds. It will be modelled as a shifted log-normal, so parameter estimations and inferential tests are conducted on values expected to fall in the range [-3, 0], [best, worst].
Story recall - immediate recall | Six months follow-up
  This is an "ecologically valid" test of short term memory. A story with 25 semantic units is read aloud and the participant re-tells the story immediately. The score is the number of items correctly recalled, i.e., 0 to 25.
  Two stories were used; one was read aloud as usual. The other was read aloud while a radio program was playing in the background.
  Range of outcome: 0 (worst) to 25 (best).
Working memory | Six months follow-up
  Subjective experience of working memory is assessed using the Working Memory Questionnaire (Vallat-Azouvi, Pradat-Diehl, & Azouvi, 2012). A global score, and three subscales (attention, storage and executive) is computed as mean sumscores.
  Range of outcome: 0 (not at all a problem, best) to 4 (Extremely a problem, worst)
  Range of outcome:
Brain injury symptoms | Six months follow-up
  Brain injury symptoms assessed by close relatives, were derived from the European Brain Injury Questionnaire (EBIQ). Eight subscales were calculated by mean sumscores:
  "Core": global brain injury symptomatology (32 items) "Somatic" (7 items) "Cognition" (11 items) "Impulsivity" (10 items) "Depression" (5 items) "Communication" (4 items) "Difficulties in social interactions" (5 items) "Fatigue" (8 items). Outcome range: From 0 ("not at all", best) to 2 ("a lot", worst).
Fatigue | Six months follow-up
  Fatigue is assessed using the Mental Fatigue Scale sum score (Birgitta Johansson, Starmark, Berglund, Rödholm, & Rönnbäck, 2010).
  A total of 14 items are scored as a sumscore and values above 10.5 are considered problematic.
  Outcome range: 0 (best) to 42 (worst).
Stress, Anxiety, and Depression | Six months follow-up
  Stress, Anxiety, and depression is assessed using the sum scores of the three individual scales of the Depression Anxiety Stress Scales questionnaire (Lovibond & Lovibond, 1995). Each subscale contains 7 items scored from 0-3. To get the final scores the sumscores are multiplied by 2.
  Range of outcome (stress): 0 (best) to 42 (worst) Range of outcome (anxiety): 0 (best) to 42 (worst) Range of outcome (depression): 0 (best) to 42 (worst)
Functioning | 6 months follow-up
  Functioning is assessed using the Impact on Participation and Autonomy questionnaire (Cardol, Haan, Bos, Jong, & Groot, 1999). Three subscales were used (Family, Social, and work scale) containing 7, 7 and 6 items respectively.
  Outcome range: each item is scored between 0 (very poor, worst) to 4 (very good, best). Sumscores are calculated and dichotomized by the 50th percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas K Lindeløv, Principal Investigator — Department for Communication and Psychology, Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindelov JK, Overgaard R, Overgaard M. Improving working memory performance in brain-injured patients using hypnotic suggestion. Brain. 2017 Apr 1;140(4):1100-1106. doi: 10.1093/brain/awx001. PMID 28335012
- [Background] Milos R. Hypnotic exploration of amnesia after cerebral injuries. Int J Clin Exp Hypn. 1975 Apr;23(2):103-10. doi: 10.1080/00207147508415934. No abstract available. PMID 1120625
- [Background] Sullivan DS, Johnson A, Bratkovitch J. Reduction of behavioral deficit in organic brain damage by use of hypnosis. J Clin Psychol. 1974 Jan;30(1):96-8. doi: 10.1002/1097-4679(197401)30:13.0.co;2-a. No abstract available. PMID 4811938
- [Background] Kihlstrom JF, Glisky ML, McGovern S, Rapcsak SZ, Mennemeier MS. Hypnosis in the right hemisphere. Cortex. 2013 Feb;49(2):393-9. doi: 10.1016/j.cortex.2012.04.018. Epub 2012 May 15. PMID 22705266
- [Background] Laidlaw TM. Hypnosis and attention deficits after closed head injury. Int J Clin Exp Hypn. 1993 Apr;41(2):97-111. doi: 10.1080/00207149308414541. PMID 8468107
- [Background] Cedercreutz C, Lahteenmaki R, Tulikoura J. Hypnotic treatment of headache and vertigo in skull injured patients. Int J Clin Exp Hypn. 1976 Jul;24(3):195-201. doi: 10.1080/00207147608416201. No abstract available. PMID 1262079
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839